CLINICAL TRIAL: NCT00355121
Title: Immunogenicity and Safety of Meningococcal (Serogroups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Children Aged 4 to 6 Years in the US When Administered Concomitantly With a Fifth Dose Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed.
Brief Title: Study of Menactra® in Children Aged 4 to 6 Years When Administered Concomitantly With a Fifth Dose of DAPTACEL®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTA43
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Meningococcal Meningitis; Tetanus; Diphtheria; Pertussis; Poliomyelitis
Keywords: Meningococcal meningitis; Tetanus; Diphtheria; Pertussis; Poliomyelitis; Neisseria meningitidis
MeSH Terms: conditions — Meningitis, Meningococcal; Tetanus; Diphtheria; Whooping Cough; Poliomyelitis | interventions — Haemophilus influenzae type b-polysaccharide vaccine-diphtheria toxoid conjugate; Meningococcal Vaccines; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): DAPTACEL® + IPOL on Day 0 and Menactra on Day 30
  Interventions: Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Group 2 (Experimental): DAPTACEL® + Menactra® on Day 0 and IPOL on Day 30
  Interventions: Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine
- Group 3 (Experimental): Menactra® + IPOL on Day 0 and DAPTACEL® on Day 30
  Interventions: Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL IM of each vaccine. (DAPTACEL® + IPOL on Day 0 and Menactra on Day 30)
  Other Names: Menactra®; DAPTACEL®; IPOL
  Arms: Group 1
Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, IM of each vaccine. (DAPTACEL® + Menactra® on Day 0 and IPOL on Day 30)
  Other Names: Menactra®; DAPTACEL®; IPOL
  Arms: Group 2
Biological: Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, IM of each vaccine (Menactra® + IPOL on Day 0 and DAPTACEL® on Day 30)
  Other Names: Menactra®; DAPTACEL®; IPOL
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the concomitant administration of Menactra® vaccine and DAPTACEL® vaccine.

The main objectives are:

Immunogenicity:

To evaluate the antibody responses to both vaccines when Menactra vaccine is given concomitantly with DAPTACEL® compared to when either vaccine is given alone.

Safety:

To evaluate the rate of local and systemic reactions when DAPTACEL® and Menactra vaccines are administered concomitantly compared to when each vaccine is given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by medical history and physical examination.
* Aged 4 to < 7 years at the time of study vaccination on Day 0.
* Informed consent form that has been approved by the Institutional Review Board (IRB) and signed/dated by the parent or legal guardian.
* Previous documented vaccination history of 4th dose diphtheria, tetanus and acellular pertussis (DTaP) series.

Exclusion Criteria:

* Serious chronic disease (e.g. cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, hematologic)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within the last 72 hours or temperature ≥ 100.4°F (≥ 38°C) at the time of enrollment
* History of documented invasive meningococcal disease or previous meningococcal vaccination
* Received a 5th dose vaccination with any tetanus, diphtheria or pertussis vaccine, or 4th dose of IPV prior to this study.
* Received either immune globulin or other blood products within the last 3 months; or received injected or oral corticosteroids, or other immunomodulator therapy, within 6 weeks of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting < 7 days and individuals (e.g., asthmatics) on a short schedule of oral steroids lasting 3 to 4 days may be included in the trial as long as they have not received more than one course within the last 2 weeks prior to enrollment.
* Received oral or injected antibiotic therapy within the 72 hours prior to any blood draw.
* Suspected or known hypersensitivity to any of the study vaccine components, history of serious or life-threatening reaction to the trial vaccines or a vaccine containing the same substances.
* Thrombocytopenia or a bleeding disorder contraindicating IM vaccination.
* Unavailable for the entire study period, or unable to attend the scheduled visits or to comply with the study procedures.
* Enrolled in another clinical trial.
* Diagnosed with any condition, which, in the opinion of the physician investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Received any other vaccine 30 days prior to the first study vaccination or scheduled to receive any vaccination during the course of the study.
* Personal or family history of Guillain-Barré Syndrome (GBS).

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 882 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (26):
- United States (26):
  - Little Rock, Arkansas
  - Boulder, Colorado
  - Atlanta, Georgia
  - Layton, UT 84041, Georgia
  - Bardstown, Kentucky
  - Woburn, Massachusetts
  - Bridgeton, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Rochester, New York
  - Syracuse, New York
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - University Heights, Ohio
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Layton, Utah
  - Ogden, Utah
  - Pleasant Grove, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Norfolk, Virginia
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 October 2006 to 21 June 2007 in 45 medical centers in the US.
Pre-assignment Details: A total of 881 participants who met the inclusion and exclusion criteria were enrolled. Data on 879 that were vaccinated are presented in this reported.
Groups:
- Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30: Participants who received single doses of diphtheria and tetanus toxoids and acellular pertussis vaccine adsorbed (DAPTACEL) and poliovirus vaccine inactivated (IPOL) at Visit 1 and a single dose of meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) at Visit 2
- Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30: Participants who received single doses of diphtheria and tetanus toxoids and acellular pertussis vaccine adsorbed (DAPTACEL) and meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) at Visit 1 and a single dose of poliovirus vaccine inactivated (IPOL) at Visit 2
- Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30: Participants who received single doses of meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) diphtheria and poliovirus vaccine inactivated (IPOL) tetanus toxoids at Visit 1 and a single dose of acellular pertussis vaccine adsorbed (DAPTACEL) at Visit 2
Period: Overall Study
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Started | 353 | 353 | 175
Completed | 332 | 324 | 170
Not Completed | 21 | 29 | 5
Not completed — Did not receive study vaccine | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 7 | 9 | 1
Not completed — Lost to Follow-up | 4 | 7 | 1
Not completed — Withdrawal by Subject | 9 | 10 | 2
Not completed — Serious adverse events | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30 | Total
Number analyzed (Participants) | 353 | 353 | 175 | 881
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 353 | 353 | 175 | 881
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 4.5 (0.48) | 4.5 (0.51) | 4.5 (0.49) | 4.5 (0.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 182 | 73 | 427
  Male | 181 | 171 | 102 | 454
Region of Enrollment [Number; unit: participants]
  United States | 353 | 353 | 175 | 881

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibodies Against Diphtheria and Tetanus at ≥ 1.0 IU/mL After DAPTACEL Vaccination
Description: Serum antibody titers were assessed for diphtheria by a seroneutralization assay and for tetanus by enzyme linked immunosorbent assay.
Time Frame: Day 30 post-vaccination (Visit 1)
Population: Serum antibody titers were assessed in the per-protocol population. (Participants in Group 3 did not receive DAPTACEL vaccine at Visit 1)
Measure: Number; unit: Participants
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 250 | 238 | 0
Participants
  Diphtheria Antibody Concentration ≥ 1.0 IU/mL | 249 | 238 |
  Tetanus Antibody Concentration ≥ 1.0 IU/mL | 246 | 236 |

2. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W-135 After Menactra Vaccination at Visit 1.
Description: Serum antibody titers against meningococcal serogroups A, C, Y, and W-135 were assessed by serum bactericidal assay using human complement (SBA HC)
Time Frame: Day 30 post-vaccination (Visit 1)
Population: Serum antibody titers were assessed in the per-protocol population. (Participants in Group 1 did not receive Menactra vaccine at Visit 1)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 0 | 238 | 121
Titers
  Serogroup A (N = 0, 131, 104) |  | 10.8 [8.7 to 13.3] | 10.4 [8.1 to 13.3]
  Serogroup C (N = 0, 131, 103) |  | 8.1 [6.3 to 10.5] | 7.8 [5.8 to 10.7]
  Serogroup Y (N = 0, 131, 104) |  | 18.1 [14.2 to 22.9] | 26.2 [20.0 to 34.4]
  Serogroup W-135 (N = 0, 131, 104) |  | 22.8 [18.5 to 28.1] | 21.7 [16.6 to 28.4]

3. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies Against the Pertussis Antigens After DAPTACEL Vaccination at Visit 1
Description: Serum antibody titers against pertussis were assessed for pertussis toxoid (PT), filamentous hemagglutinin (FHA), Fimbriae types 2 and 3 (FIM), and pertactin (RN) by enzyme linked immunosorbent assay (ELISA).
Time Frame: Day 30 post-vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 250 | 238 | 0
EU/mL
  Pertussis toxoid (PT; N = 243, 236, 0) | 70.0 [63.0 to 77.8] | 71.0 [63.8 to 79.0] |
  Filamentous hemagglutinin (FHA; N = 246, 237, 0) | 133 [117 to 152] | 145 [127 to 165] |
  Fimbriae Types 2 and 3 (FIM; N = 243, 238, 0) | 123 [92.5 to 164] | 113 [84.0 to 151] |
  Pertactin (PRN; N = 247, 238, 0) | 115 [97.0 to 136] | 118 [102 to 137] |

4. Secondary Outcome: Serum Bactericidal Assay Using Human Complement Geometric Mean Titers for Serogroups A, C, Y, and W-135 After Menactra Vaccination
Description: as for outcome 2
Time Frame: Day 30 post-vaccination
Population: Serum antibody titers were assessed in the per protocol population. Participants in Group 1 received Menactra vaccine at Visit 2, Group 3 at Visit 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 250 | 0 | 121
Titers
  Serogroup A (N = 137, 0, 104) | 6.7 [5.7 to 8.0] |  | 10.4 [8.1 to 13.3]
  Serogroup C (N = 138, 0, 103) | 3.3 [2.7 to 3.9] |  | 7.8 [5.8 to 10.7]
  Serogroup Y (N = 138, 0, 104) | 6.5 [5.1 to 8.2] |  | 26.2 [20.0 to 34.4]
  Serogroup W-135 (N = 138, 0, 104) | 8.4 [6.7 to 10.6] |  | 21.7 [16.6 to 28.4]

5. Secondary Outcome: Number of Participants Reporting Fever When DAPTACEL and Menactra Vaccines Were Administered Concomitantly and Those Reporting When DAPTACEL Was Administered With IPOL Vaccine
Description: Fever was defined as a maximum oral temperature of ≥ 100.4ºF.
Time Frame: Day 0 through Day 7 post-vaccination at Visit 1
Population: Safety analysis was on enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 341 | 344 | 0
Participants | 27 | 18 |

6. Other Pre Specified Outcome: Geometric Mean Titers Against Poliovirus After IPOL Vaccination.
Description: Serum antibodies were assessed for poliovirus types 1, 2, and 3 by serum neutralization assay.
Time Frame: Day 30 post-vaccination
Population: Serum antibody titers were assessed in the per-protocol population. (Participants received IPOL at Visit 1 in Group 1 and 3, and at Visit 2 for Group 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 250 | 238 | 121
Titers
  Type 1 (N = 243, 235, 120) | 5094.8 [4427.8 to 5862.4] | 5767 [4982.7 to 6674.9] | 4885.1 [4013.2 to 5946.4]
  Type 2 (N = 245, 237, 120) | 5209.5 [4549.0 to 5966.0] | 6195.6 [5325.3 to 7208.1] | 5373.6 [4461.0 to 6472.8]
  Type 3 (N = 245, 236, 120) | 6777.5 [5766.9 to 7965.2] | 7815.9 [6601.0 to 9254.5] | 5843 [4523.4 to 7547.6]

7. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions After Vaccinations at Visit 1
Description: Solicited Injection Site Reactions: Pain, Erythema, and Redness. Solicited Systemic Reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
Time Frame: Day 0 through Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Number analyzed (Participants) | 341 | 344 | 169
Participants
  Any Injection Site Pain: DAPTACEL | 236 | 229 | NA — DAPTACEL was not administered at Visit 1
  Grade 3 Pain (Incapacitating): DAPTACEL | 2 | 2 | NA — DAPTACEL was not administered at Visit 1
  Any Injection Site Erythema: DAPTACEL | 161 | 161 | NA — DAPTACEL was not administered at Visit 1
  Grade 3 Erythema (≥ 2 in): DAPTACEL | 75 | 73 | NA — DAPTACEL was not administered at Visit 1
  Any Injection Site Swelling: DAPTACEL | 113 | 109 | NA — DAPTACEL was not administered at Visit 1
  Grade 3 Swelling (≥ 2 in): DAPTACEL | 54 | 41 | NA — DAPTACEL was not administered at Visit 1
  Any Injection Site Pain: Menactra | NA — Menactra was not administered at Visit 1 | 201 | 93
  Grade 3 Pain (Incapacitating): Menactra | NA — Menactra was not administered at Visit 1 | 1 | 2
  Any Injection Site Erythema: Menactra | NA — Menactra was not administered at Visit 1 | 103 | 31
  Grade 3 Erythema (≥ 2 in): Menactra | NA — Menactra was not administered at Visit 1 | 16 | 6
  Any Injection Site Swelling: Menactra | NA — Menactra was not administered at Visit 1 | 66 | 21
  Grade 3 Swelling (≥ 2 in): Menactra | NA — Menactra was not administered at Visit 1 | 18 | 5
  Any Injection Site Pain: IPOL | 207 | NA — IPOL was not administered at Visit 1 | 98
  Grade 3 Pain (Incapacitating): IPOL | 3 | NA — IPOL was not administered at Visit 1 | 2
  Any Injection Site Erythema: IPOL | 59 | NA — IPOL was not administered at Visit 1 | 23
  Grade 3 Erythema (≥ 2 in): IPOL | 10 | NA — IPOL was not administered at Visit 1 | 2
  Any Injection Site Swelling: IPOL | 39 | NA — IPOL was not administered at Visit 1 | 12
  Grade 3 Swelling (≥ 2 in): IPOL | 8 | NA — IPOL was not administered at Visit 1 | 2
  Any Fever | 27 | 18 | 13
  Grade 3 Fever (> 39.5 ºC or ≥ 103.2 ºF) | 1 | 3 | 0
  Any Headache | 48 | 42 | 22
  Grade 3 Headache (Prevents daily activities) | 2 | 1 | 0
  Any Malaise | 86 | 81 | 44
  Grade 3 Malaise (Prevents daily activities) | 8 | 2 | 5
  Any Myalgia | 153 | 123 | 44
  Grade 3 Myalgia (Prevents daily activities) | 6 | 3 | 0

8. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions After Vaccination at Visit 2
Description: as for outcome 7
Time Frame: Day 0 through Day 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Groups:
- Group 1: Menactra on Day 30 (Visit 2): Participants who received single doses of diphtheria and tetanus toxoids and acellular pertussis vaccine adsorbed (DAPTACEL) and poliovirus vaccine inactivated (IPOL) at Visit 1 and a single dose of meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) at Visit 2
- Group 2: IPOL on Day 30 (Visit 2): Participants who received single doses of diphtheria and tetanus toxoids and acellular pertussis vaccine adsorbed (DAPTACEL) and meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) at Visit 1 and a single dose of poliovirus vaccine inactivated (IPOL) at Visit 2
- Group 3: DAPTACEL on Day 30 (Visit 2): Participants who received single doses of meningococcal polysaccharide diphtheria toxoid conjugate vaccine (Menactra) diphtheria and poliovirus vaccine inactivated (IPOL) tetanus toxoids at Visit 1 and a single dose of acellular pertussis vaccine adsorbed (DAPTACEL) at Visit 2
Arm/Group | Group 1: Menactra on Day 30 (Visit 2) | Group 2: IPOL on Day 30 (Visit 2) | Group 3: DAPTACEL on Day 30 (Visit 2)
Number analyzed (Participants) | 328 | 327 | 165
Participants
  Any Injection Site Pain | 168 | 128 | 85
  Grade 3 Pain (Incapacitating) | 2 | 1 | 0
  Any Injection Site Erythema | 80 | 54 | 42
  Grade 3 Erythema (≥ 2 inches) | 24 | 2 | 18
  Any Injection Site Swelling | 58 | 31 | 32
  Grade 3 Swelling (≥ 2 inches) | 19 | 1 | 10
  Any Fever | 12 | 17 | 11
  Grade 3 Fever (> 39.5 ºC or ≥ 103.2 ºF) | 1 | 1 | 0
  Any Headache | 27 | 21 | 12
  Grade 3 Headache (Prevents daily activities) | 1 | 2 | 1
  Any Malaise | 46 | 47 | 37
  Grade 3 Malaise (Prevents daily activities) | 4 | 8 | 3
  Any Myalgia | 78 | 55 | 42
  Grade 3 Myalgia (Prevents daily activities) | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination for up to 6 months post-vaccination at Visit 2.
Arm/Group | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30
Serious Adverse Events (participants affected / at risk) | 0/341 | 2/344 | 1/169
Other Adverse Events (participants affected / at risk) | 236/341 | 229/344 | 98/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 (N=341) | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 (N=344) | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30 (N=169)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: DAPTACEL + IPOL on Day 0 / Menactra on Day 30 (N=341) | Group 2: DAPTACEL + Menactra on Day 0 / IPOL on Day 30 (N=344) | Group 3: Menactra + IPOL on Day 0 / DAPTACEL on Day 30 (N=169)
Injection Site Pain (General disorders) | 236/329 (236) | 229/330 (229) | 98/166 (98)
Injection Site Erythema (General disorders) | 161/330 (161) | 161/330 (161) | 42/163 (42)
Injection Site Swelling (General disorders) | 113/330 (113) | 109/329 (109) | 32/162 (32)
Fever (General disorders) | 27/328 (27) | 18/325 (18) | 13/163 (13)
Malaise (General disorders) | 86/331 (86) | 81/330 (81) | 44/165 (44)
Myalgia (Musculoskeletal and connective tissue disorders) | 153/331 (153) | 123/330 (123) | 44/165 (44)
Headache (Nervous system disorders) | 48/331 (48) | 42/330 (42) | 22/165 (22)
Vomiting (Gastrointestinal disorders) | 14 (14) | 18 (18) | 10 (10)
Injection Site Induration (General disorders) | 22 (22) | 16 (16) | 12 (12)
Injection Site Pruritus (General disorders) | 18 (18) | 15 (15) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (38) | 39/343 (39) | 23 (23)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 22/343 (22) | 9 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 12/343 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications